CLINICAL TRIAL: NCT00895661
Title: Phase II Trial of Increased Dose Rituximab Plus Maintenance Rituximab for Initial Systemic Treatment of Indolent B-Cell Lymphomas
Brief Title: High Dose Rituximab for Initial Treatment of Indolent B-Cell Lymphomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Jeremy Abramson, MD, Director, Lymphoma Program, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-054
Record Dates: First submitted 2009-05-06; First posted 2009-05-08 (Estimated); Results first posted 2017-05-09 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-05

CONDITIONS: B-cell Lymphoma; Indolent B-cell Lymphoma
Keywords: rituximab
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rituximab (Other): single-arm, open-label, interventional
  Interventions: Drug: rituximab

INTERVENTIONS:
Drug: rituximab — Increased dose (750 mg/m2) intravenously for 4 weekly doses followed by maintenance dosing once every three months for up to 2 years. Maintenance dose is standard (375 mg/m2).
  Other Names: Rituxan

SUMMARY:
The purpose of this clinical trial is to see if increased doses of rituximab are safe and effective for the initial treatment of indolent B-cell lymphomas. Rituximab (Rituxan) is a type of drug called an "antibody" that specifically targets B-cell lymphoma cells, and is approved by the FDA for the treatment of indolent B-cell non-hodgkin lymphomas and certain other types of non-hodgkin lymphomas. Standard doses currently used may not be achieving maximal efficacy. Higher doses have been shown to be safe in other clinical trials, and may offer superior efficacy to the current standard dose. This trial also employs intermittent maintenance doses of rituximab at the standard dose, which has been shown to prolong remissions and survival in patients with relapsed indolent B-cell lymphomas. This trial is designed to show that higher dose rituximab plus maintenance rituximab can achieve similarly good results to chemotherapy approaches, but without chemotherapy-related toxicity.

DETAILED DESCRIPTION:
* All participants will receive increased-dose rituximab through a vein in the arm once a week for 4 weeks (on Days 1, 8, 15, and 22 of the initial 28-day study cycle). This first cycle of study treatment is called the Induction Phase. If the participant responds well to the Induction Phase, they then may continue to the Maintenance Therapy Phase, where they will receive a lower dose of rituximab once every three months for up to 2 years.
* During the Induction Phase, the following procedures will take place before the participant receives each dose of rituximab: medical review, physical exam, performance status, and ECG. Blood tests will be drawn about 30-60 minutes after the first dose of rituximab on Day 1. Samples will be drawn immediately before each dose and again 30-60 minutes after each dose on Days 1, 8, 15 and 22.
* During the Maintenance Therapy Phase, the following procedures will take place before the participant receives each dose of rituximab: medical review, physical exam, performance status, ECG, blood tests and response assessments by CT scan.

ELIGIBILITY:
Inclusion Criteria:

* Indolent B-Cell NHL of the following histologies:

  1. Follicular lymphoma (grades 1-3A);
  2. marginal zone lymphoma (extranodal, nodal or splenic):

     * Extranodal marginal zone lymphomas (MALT lymphomas) may not be candidates for cure with antibiotics or local radiotherapy. Patients who have failed antibiotics or local therapy are eligible for the protocol as long as they have measurable disease and are naive to chemotherapy and monoclonal antibody;
     * splenic marginal zone lymphoma patients may have received prior splenectomy as long as they have measureable disease and are naive to chemotherapy and monoclonal antibody therapy;
  3. Small lymphocytic lymphoma (must have less than 5000 circulating clonal B-lymphocytes);
  4. Indolent CD20+ B-cell lymphoma not otherwise specified with CD20+ expression
* Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as 20mm or greater with conventional techniques or as 10mm or greater with spiral CT scan
* No previous chemotherapy, antibody therapy or radioimmunotherapy for NHL. Patients previously treated with external bean radiation alone, surgery, or with antibiotics are eligible
* 18 years of age or older
* Life expectancy of greater than 3 months
* ECOG performance status of 2 or less
* Adequate bone marrow function
* Use of adequate contraception

Exclusion Criteria:

* Prior chemotherapy, monoclonal antibody therapy or radioimmunotherapy for lymphoma
* Receiving any other investigational agent
* Known brain metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to rituximab
* HIV positivity
* Active hepatitis B infection
* Candidate for curative radiotherapy, unless radiation therapy is considered too toxic (as in abdominal disease), or is refused by the patient
* NYHA Classification III or IV disease
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection that is not optimally treated with antibiotics, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women
* Individuals with a history of a different malignancy except for the following circumstances:

  1. disease-free for at least 1 year and are deemed by the investigator to be at low risk for recurrence of that malignancy;
  2. localized prostate cancer, prostate cancer with elevated PSA but no measurable disease on CT scans or bone scan, cervical cancer in situ; and
  3. non-melanoma skin cancers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2010-10 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Abramson, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rituximab
Started | 40
Completed | 37
Not Completed | 3
Not completed — Death | 1
Not completed — reason unknown | 2

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: years] | 60 [36 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 40
Lymphoma type [Count of Participants; unit: Participants]
  Follicular | 31
  Marginal zone | 4
  Small lymphocytic | 3
  Indolent B cell, not otherwise specified | 2
Involvement of >4 nodal sites [Count of Participants; unit: Participants] | 17
Hgb<12 g/dL [Count of Participants; unit: Participants] | 9
elevated LDH (Lactate dehydrogenase) [Count of Participants; unit: Participants] | 11
Follicular lymphoma prognostic index (FLIPI) [Count of Participants; unit: Participants]
  Low risk | 6
  Intermediate risk | 15
  High risk | 17
  FLIPI score not available | 2

OUTCOME MEASURES:

1. Primary Outcome: Determine Complete Response Rate (CRR) of Increased Dose Rituximab in Indolent B-cell Lymphomas
Description: CR requires all of the following:
  1. Regression to normal size on CT (≤ 1.5 cm in their greatest transverse diameter for nodes ≥ 1.5 cm before therapy). Previously involved nodes that were 1.1 to 1.5 cm in their greatest transverse diameter before treatment must have decreased to <1 cm in their greatest transverse diameter after treatment, or by more than 75% in the sum of the products of the greatest diameters (SPD).
  2. The spleen, if considered to be enlarged before therapy on the basis of a CT scan, must have regressed in size and must not be palpable on physical examination.
  3. If bone marrow is known to be involved at the beginning, then repeat biopsy documents clearance
Time Frame: after a median number of 8 maintenance cycles, up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab
Number analyzed (Participants) | 40
Participants | 21

2. Secondary Outcome: Overall Response Rate (ORR)
Description: Complete Response (CR): see definition in primary outcome
  Partial Response (PR):
  1. ≥50% decrease in SPD of up to 6 largest dominant masses
  2. No new sites of disease or increase in the size of the other nodes, liver, or spleen.
  3. Splenic and hepatic nodules must regress by at least 50% in the SPD.
  Overall Response (OR) = CR + PR.
Time Frame: after a median number of 8 maintenance cycles, up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab
Number analyzed (Participants) | 40
Participants | 32

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Progressive Disease (PD) or Relapsed Disease (RD):
  1. Appearance of a new lesion(s) > 1.5 cm in any axis, ≥ 50% increase in SPD of more than one node, or ≥50% increase in longest diameter of a previously identified node > 1 cm in short axis.
  2. >50% increase from nadir in the SPD of any previous lesions PFS is number of participants who have not died or had PD or RD.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab
Number analyzed (Participants) | 40
Participants | 19

4. Secondary Outcome: Incidence of Severity of Infusion Reactions, Infections and Neutropenia
Description: Toxicity grades: 1 = mild, 2 = moderate, 3 = severe, 4 = life-threatening
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab
Number analyzed (Participants) | 40
Participants
  Grade 3/4 neutropenia | 3
  Any allergic reactions with infusions | 19
  Grade 3 allergic reactions with infusions | 2

ADVERSE EVENTS:
Arm/Group | Rituximab
Serious Adverse Events (participants affected / at risk) | 4/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab (N=40)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) — grade 3, unexpected and unrelated
Small bowel obstruction (Gastrointestinal disorders) | 1 (1) — grade 4, unexpected and unrelated
Cellulitis (toe) (Infections and infestations) | 1 (1) — grade 3, expected and possibly related
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — grade 3, unexpected and possibly related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab (N=40)
Neutrophils (Blood and lymphatic system disorders) | 40 (495)
Allergic reaction (Immune system disorders) | 40 (493)
Infection-other (Infections and infestations) | 40 (493)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 40 (493)
Fatigue (General disorders) | 24 (97)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (34)
Hyperglycemia (Metabolism and nutrition disorders) | 14 (52)
Hemoglobin (Blood and lymphatic system disorders) | 13 (38)
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 11 (32)
Leukocytes (Blood and lymphatic system disorders) | 11 (32)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 10 (19)
Infection Gr0-2 neut- upper airway (Infections and infestations) | 10 (14)
Fever w/o neutropenia (General disorders) | 10 (12)
Abdomen- pain (General disorders) | 9 (21)
Nausea (Gastrointestinal disorders) | 9 (21)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (19)
Dizziness (Nervous system disorders) | 8 (21)
Allergic rhinitis (Immune system disorders) | 8 (20)
Head/headache (General disorders) | 8 (20)
Sweating (General disorders) | 8 (19)
Skin-other (Skin and subcutaneous tissue disorders) | 8 (16)
Back-pain (General disorders) | 8 (10)
Lymphopenia (Blood and lymphatic system disorders) | 7 (15)
Pain-other (General disorders) | 7 (11)
Insomnia (General disorders) | 6 (27)
Pelvic-pain (General disorders) | 6 (15)
Joint-pain (General disorders) | 6 (14)
Anxiety (Nervous system disorders) | 5 (18)
Anorexia (Gastrointestinal disorders) | 5 (13)
AST- SGOT (Metabolism and nutrition disorders) | 5 (8)
Dyspepsia (Gastrointestinal disorders) | 5 (7)
Platelets (Blood and lymphatic system disorders) | 5 (6)
Infection Gr0-2 neut- bronchus (Infections and infestations) | 5 (5)
Rigors/chills (General disorders) | 5 (5)
Neuropathy-sensory (Nervous system disorders) | 4 (18)
Alkaline phosphatase (Metabolism and nutrition disorders) | 4 (13)
ALT- SGPT (Metabolism and nutrition disorders) | 4 (10)
Extremity-limb- pain (General disorders) | 4 (10)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 4 (9)
Infection Gr0-2 neut- sinus (Infections and infestations) | 4 (6)
Neck- pain (General disorders) | 4 (6)
Vomiting (Gastrointestinal disorders) | 4 (6)
Hyperuricemia (Metabolism and nutrition disorders) | 3 (9)
Urinary frequency/urgency (Renal and urinary disorders) | 3 (8)
Constipation (Gastrointestinal disorders) | 3 (7)
Creatinine (Metabolism and nutrition disorders) | 3 (6)
GI-other (Gastrointestinal disorders) | 3 (6)
Hearing-other (Ear and labyrinth disorders) | 3 (6)
Edema head and neck (Blood and lymphatic system disorders) | 3 (5)
Hematologic-other (Blood and lymphatic system disorders) | 3 (5)
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Bronchospasm- wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Chest/thoracic pain NOS (General disorders) | 3 (4)
Muscle- pain (General disorders) | 3 (4)
Flu-like syndrome (General disorders) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 3 (3)
Palpitations (Cardiac disorders) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (9)
Sinus bradycardia (Cardiac disorders) | 2 (9)
Dysphagia (Gastrointestinal disorders) | 2 (8)
Sinus tachycardia (Cardiac disorders) | 2 (7)
Cholecystitis (Hepatobiliary disorders) | 2 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (5)
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 2 (5)
Dry mouth (Gastrointestinal disorders) | 2 (3)
Esophagitis (Gastrointestinal disorders) | 2 (3)
Hyopthyroidism (Endocrine disorders) | 2 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (3)
Infection Gr0-2 neut- skin (Infections and infestations) | 2 (3)
Infection Gr0-2 neut- urinary tract (Infections and infestations) | 2 (3)
Otitis- middle ear (non-infectious) (Ear and labyrinth disorders) | 2 (3)
Taste disturbance (Gastrointestinal disorders) | 2 (3)
Chest wall- pain (General disorders) | 2 (2)
Dehydration (Gastrointestinal disorders) | 2 (2)
Edema limb (Blood and lymphatic system disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Infection Gr0-2 neut- lung (Infections and infestations) | 2 (2)
Metabolic/Laboratory-other (Metabolism and nutrition disorders) | 2 (2)
Ocular-other (Eye disorders) | 2 (2)
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Weight gain (General disorders) | 2 (2)
Weight loss (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No